CLINICAL TRIAL: NCT05482282
Title: Comparison of Immunogenicity and Safety of DTP-HB-Hib Using New Hepatitis B Bulk (Bio Farma) With Pentabio® Vaccine Primed With Recombinant Hepatitis B at Birth Dose Using New Hepatitis B Bulk (Bio Farma), in Indonesian Infants
Brief Title: Immunogenicity and Safety of DTP-HB-Hib Using New Hepatitis B Bulk (Bio Farma)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: The products will be replace with others.
Sponsor: PT Bio Farma (Industry)
Collaborators: Hasan Sadikin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Penta BS22
Record Dates: First submitted 2022-07-29; First posted 2022-08-01 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: Diphtheria Vaccine Adverse Reaction; Tetanus Vaccine Adverse Reaction; Pertussis Vaccine Adverse Reaction; Haemophilus Influenzae Type B Vaccine Adverse Reaction; Hepatitis B Vaccine Adverse Reaction
Keywords: DTP-HB-Hib Vaccine; Hepatitis B Vaccine
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Vaccines

STUDY DESIGN:
Intervention Model Description: Subjects neonates: Randomized, double blind, 2 arms parallel groups, prospective intervention study
Who Masked: Participant, Investigator
Masking Description: Double (Participant, Investigator) Observer Blind : Investigational Product and Active Comparator are masking Lot number is masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Recombinant Hep B new Bulk + Penta with Recombinant HepB new Bulk (Experimental): 1 dose Recombinant Hepatitis B new Bulk vaccine at birth + 3 doses Pentavalent with Recombinant HepB new Bulk vaccine
  Interventions: Biological: Recombinant Hepatitis B new Bulk vaccine; Biological: DTP-HB-Hib with Recombinant Hepatitis B new Bulk vaccine
- Hep B (Registered) + Pentabio (Registered) (Active Comparator): 1 dose Recombinant Hepatitis B vaccine (Registered) + 3 doses Pentabio with Recombinant HepB new Bulk vaccine
  Interventions: Biological: Recombinant Hepatitis B vaccine (Registered BioFarma); Biological: Pentabio

INTERVENTIONS:
Biological: Recombinant Hepatitis B new Bulk vaccine — 1 dose of Recombinant Hepatitis B vaccine using new Hepatitis B bulk (Bio Farma)
  1 dose of 0.5 ml Recombinant Hepatitis B new Bulk vaccine dose of DTP-HB-Hib using new Hepatitis B Bulk vaccine injected intramuscularly into the left external antero-lateral thigh region.
  Arms: Recombinant Hep B new Bulk + Penta with Recombinant HepB new Bulk
Biological: DTP-HB-Hib with Recombinant Hepatitis B new Bulk vaccine — 3 doses of DTP-HB-Hib with Recombinant Hepatitis B new Bulk vaccine
  Arms: Recombinant Hep B new Bulk + Penta with Recombinant HepB new Bulk
Biological: Recombinant Hepatitis B vaccine (Registered BioFarma) — 1 dose of Recombinant Hepatitis B vaccine (Registered Bio Farma)
  Arms: Hep B (Registered) + Pentabio (Registered)
Biological: Pentabio — 3 doses of Pentabio
  Arms: Hep B (Registered) + Pentabio (Registered)

SUMMARY:
This bridging study is a randomized, double-blind, two arms parallel group, prospective intervention study. The primary objective of this study is to evaluate protectivity of DTP-HB-Hib Vaccine (Bio Farma) using new Hepatitis B bulk (Bio Farma).

DETAILED DESCRIPTION:
This bridging study is a randomized, double blind, two arms parallel groups, prospective intervention study. Total 220 infants, 0-3 days old will be involved in this study. The subject will be divided into 2 groups, 110 subjects are the investigational group and 110 subjects are the active comparator group.

The objective of this study is to evaluate protectivity of DTP-HB-Hib Vaccine (Bio Farma) using new Hepatitis B bulk (Bio Farma) and to asses the safety of DTP-HB-Hib Vaccine (Bio Farma) and Recombinant Hepatitis B Vaccine using new Hepatitis B bulk (Bio Farma).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, full term, newborns infants.
2. Infant born after 37-42 weeks of pregnancy.
3. Infant weighing 2500 gram or more at birth.
4. Father, mother or legally acceptable representative properly informed about the study and having signed the informed consent form.
5. Parents will commit themselves to comply with the indications of the investigator and with the schedule of the trial.

Exclusion Criteria:

1. Child concomitantly enrolled or scheduled to be enrolled in another trial.
2. Child evolving moderate or severe illness, especially infectious diseases or fever (axillary temperature 37.5 celcius degrees on Day 0).
3. Child suspected of allergy to any component of the vaccines (e.g. formaldehyde), based on anamnesis.
4. Child suspected of uncontrolled coagulopathy or blood disorders contraindicating intramuscular injection, based on anamnesis
5. Newborn suspected of congenital or acquired immunodeficiency, based on anamnesis
6. Child received or plans to receive any treatment likely to alter the immune response intravenous (immunoglobulins, blood-derived products or long term corticotherapy (> 2 weeks)).
7. Child received other vaccination with the exception of BCG and poliomyelitis.
8. Child has any abnormality or chronic disease which according to the investigator might interfere with the assessment of the trial objectives.
9. Mother with HbsAg and HIV positive (by rapid test within 30 days prior subject's birth)
10. Mother suspected of immunodeficiency disease based on anamnesis

Ages: 1 Day to 3 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
To evaluate protectivity of DTP-HB-Hib Vaccine (Bio Farma) using new Hepatitis B bulk (Bio Farma) | 28 days
  Percentage of infants with anti-diphtheria titer and anti-tetanus titer more than 0.01 IU/ml, anti HbsAg titer more than 10 mIU/ml, and anti PRP-TT titer more than 0.15 microgram/ml 28 days after the last injection of DTP-HB-Hib using new Hepatitis B bulk (Bio Farma) vaccine group.

SECONDARY OUTCOMES:
To asses the local and systemic reactions within 30 minutes | 30 minutes
  Local reaction and systemic events occurring within 30 minutes after immunization.
To asses the local and systemic reactions within 30 minutes to 7 days after immunization | 7 days
  Local reaction and systemic events occurring after 30 minutes to 7 days after immunization.
To asses the local and systemic reactions within 7 days to 28 days after immunization | 28 days
  Local reaction and systemic events occurring after 7 days to 28 days following the vaccination.
To asses the serious adverse event | 28 days
  Any serious adverse event occuring from inclusion until 28 days after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Eddy Fadlyana, MD, Principal Investigator — Hasan Sadikin General Hospital
Locations (3):
- Indonesia (3):
  - Garuda Primary Health Centre, Bandung, West Java
  - Ibrahim Adjie Primary Health Centre, Bandung, West Java
  - Puter Primary Health Centre, Bandung, West Java